CLINICAL TRIAL: NCT04548882
Title: Continued Evaluation of the Calypso Knee System for Symptom Relief in Subjects With Medial Knee Osteoarthritis, OUS
Brief Title: Calypso Knee System Clinical Sub-study, OUS Continued Evaluation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed based on continued restrictions around COVID-19
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0004
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single-arm study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Calypso Knee System (Experimental): Calypso Knee System
  Interventions: Device: Calypso Knee System

INTERVENTIONS:
Device: Calypso Knee System — The Calypso Knee System is an extra-capsular knee implant designed to fill the therapeutic gap between conservative care and more invasive surgical interventions for knee osteoarthritis.
  Other Names: Calypso System

SUMMARY:
Calypso Knee System Clinical Study, OUS for subjects with symptomatic osteoarthritis of the medial compartment of the knee. The sub-study will achieve continued evaluation of the safety and clinical effectiveness of the Calypso Knee System.

DETAILED DESCRIPTION:
This sub-study will be a single-arm, prospective, multi-center sub-study for continued evaluation of the safety and clinical effectiveness of Calypso Knee System using an additional measure of post-operative activity improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Participants age - 25 to 65 years
2. Body Mass Index (BMI) of < 35, Weight < 300 lbs
3. Knee osteoarthritis pain on the inner side of knee that has continued after at least 6 months of non-operative treatment

Exclusion Criteria:

1. Symptoms of osteoarthritis in the other knee or in lateral (outer) or patellofemoral compartments of the target knee
2. Knee ligament or meniscal instability
3. Other bone or joint conditions such as Rheumatoid arthritis, Paget's disease, Charcot's disease or general conditions such as allergy or hypersensitivity to certain metals, active infection, certain neurological conditions, use of medication such as steroids or chemotherapy that could impact study participation or results

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this pilot study is the rate of individual subject success at 24 months. A subject will be declared a clinical success if all of the following conditions are met | Change at 24 months relative to baseline
  1. Clinically Significant improvement in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Pain
  2. Clinically Significant improvement in Western Ontario and McMasters University Osteoarthritis Index (WOMAC) Function
  3. Freedom from applicable device-related SAEs requiring surgical intervention
  4. Maintenance of Implant Integrity by Radiographic Review

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kraenzlin, Study Director — Moximed